CLINICAL TRIAL: NCT04752774
Title: An Integrated Phase I/II, Multicentre, Double-blind, Randomised, Dysport and Placebo-controlled, Dose Escalation and Dose-finding Study to Evaluate the Safety and Efficacy of IPN10200 in the Treatment of Adult Upper Limb Spasticity.
Brief Title: A Study to Assess the Safety and Efficacy of IPN10200 in Adult Participants With Upper Limb Spasticity.
Acronym: LANTIMA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-FR-10200-001; 2020-003623-42 (EudraCT Number)
Record Dates: First submitted 2021-02-03; First posted 2021-02-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Spasticity
Keywords: Upper limb spasticity after stroke or traumatic brain injury
MeSH Terms: conditions — Muscle Spasticity; Brain Injuries, Traumatic | interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation (Experimental): One single administration of study medication (IPN10200, Dysport or placebo) will be injected in a dose-escalation manner. Dose-escalation will include several cohorts.
  Interventions: Biological: IPN10200; Drug: Placebo; Biological: Dysport
- Dose ranging (Experimental): Two fixed doses of IPN10200 will be administrated as a single injection into several muscle groups of the upper limb.
  Participants will be randomised in the ratio of 3:3:2 (total IPN10200 dose 1: 30 participants; total IPN10200 dose 2: 30 participants; Dysport: 20 participants)
  Interventions: Biological: IPN10200; Biological: Dysport
- Total dose (Experimental): One single injection of study medication will be administered locally into several muscle groups of the upper limb.
  Participants will be randomized in the ratio of 2:1 (Total IPN10200 dose: 30 participants; placebo: 15 participants, resulting in a total of 45 participants in Stage 3).
  Or
  Participants will be randomized in the ratio of 3:1 (IPN10200 lower dose: 30 participants; placebo: 10 participants, then IPN10200 higher dose: 30 participants; placebo: 10 participants, resulting in a total of 80 participants in Stage 3).
  Interventions: Biological: IPN10200; Drug: Placebo

INTERVENTIONS:
Biological: IPN10200 — Powder and solvent for solution for injection
Drug: Placebo — Powder and solvent for solution for injection
  Arms: Dose escalation; Total dose
Biological: Dysport — Powder for solution for injection
  Arms: Dose escalation; Dose ranging

SUMMARY:
The purpose of the study is to assess the safety and efficacy of increasing doses of IPN10200 with the aim to evaluate the Pharmacodynamics (PD) profile of IPN10200 and to establish the total IPN10200 doses(s) that offer the best efficacy/safety profile when used for the treatment of Adult upper limb (AUL) spasticity.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 70 years of age inclusive (except for dose escalation must be 18 to 65 years of age) at the time of signing the informed consent.
2. Has spastic hemiparesis following stroke or Traumatic brain injury (TBI)
3. Is at least 6 months post-stroke or TBI
4. Has never received BoNT or if previously treated, should have received their last injection of any commercialized BoNT-A or B at least 4 months prior to study Baseline
5. Has a MAS score ≥2 in the (PTMG) to be injected
6. Is eligible to receive a total recommended dose 1000 U Dysport in the upper limb when applicable.
7. Has angle of spasticity ≥5° in the PTMG to be injected.
8. Does not have any fixed contractures as defined by:

   * Complete fingers extension with Angle of arrest at slow speed (Tardieu Scale) (XV1) ≥160°
   * Complete wrist extension with XV1 ≥90°
   * Complete elbow extension with XV1 ≥160°
9. Physiotherapy, occupational therapy, splinting, use of benzodiazepine, and muscle relaxants had to be stable from at least 30 days preceding the study Baseline up to the Month 3 visit, and whenever possible until the end of the study.
10. In good health (i.e. absence of any uncontrolled systemic disease or other significant medical condition) as determined by medical history, physical and neurological examinations, clinical laboratory studies, electrocardiograms (ECGs), vital signs, and Investigator's judgment prior to randomization
11. Male and female participants Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Male participants must agree that, if their partner is at risk of becoming pregnant, they will use an effective method of contraception. The participants must agree to use the contraception during the whole period of the study.

A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: Is a woman of non-childbearing potential (WONCBP) or is a woman of childbearing potential (WOCBP) and using an acceptable contraceptive method (until the end of the study). The investigator should evaluate the potential for contraceptive method failure in relationship to the first dose of study intervention. A WOCBP must have a negative highly sensitive pregnancy test.

Exclusion Criteria:

1. Any medical condition (including severe dysphagia or airway disease) that may increase, in the opinion of the investigator, the likelihood of adverse events (AEs) related to BoNT treatment.
2. Known disease of the neuromuscular junction (e.g. Lambert-Eaton myasthenic syndrome, myasthenia gravis or amyotrophic lateral sclerosis etc.).
3. Has a history of hypersensitivity to the investigational medicinal products (or other BoNTs) or any excipient used in their formulation.
4. Clinically diagnosed significant anxiety disorder, or any other significant psychiatric disorder (e.g. depression) that might interfere with the participant's participation in the study.
5. Likely treatment with any serotype of BoNT for any condition during the study.
6. Undergone previous surgery to treat spasticity in the affected upper limb.
7. Has initiated physiotherapy within 30 days prior to Baseline (if physiotherapy initiated more than 30 days prior to Baseline and ongoing, the therapy regimen should be maintained at the same frequency and intensity throughout the study if possible or at least up to 3-months post-injection).
8. Has received previous treatment with phenol and or alcohol in the targeted upper limb any time before the study.
9. Has been treated or is likely to be treated with intrathecal baclofen during the 30 days prior to study Baseline or during the course of the study.
10. Current or planned treatment with any medications that interfere either directly or indirectly with neuromuscular transmission, such as curare-like non depolarising agents, lincosamides, polymyxins, anticholinesterases and aminoglycoside antibiotics, within 30 days prior to Baseline.
11. Use of concomitant therapy which, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study intervention, including medications affecting bleeding disorders. For patients taking vitamin K antagonists, the INR values should be controlled (between 2 and 3)
12. Currently planned or a history of tendon lengthening surgery, significant contracture or muscle atrophy at target joint or muscle in the past 6 months prior to Screening.
13. Use of any experimental device within 30 days or use of any treatment with an experimental drug within five times the documented terminal half-life of the respective drug or its metabolites or if the half-life is unknown within 30 days prior to the start of the study (prior to Baseline) and during the conduct of the study.
14. Presence of any other condition (e.g. neuromuscular disorder, muscular dystrophies, cancer cachexia, sarcopenia or other disorder that could interfere with neuromuscular function), laboratory finding or circumstance that, in the judgment of the investigator, might increase the risk to the participant or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
15. Pregnant or lactating women, or women of childbearing potential not willing to practice a highly effective form of contraception method at the beginning of the study, for the duration of the study and for the duration of the study
16. Inability to understand protocol procedures and requirements
17. Infection at the injection site(s)
18. A history of drug or alcohol abuse
19. Male participants who are not vasectomised and who have female partners of childbearing potential and are not willing to use condoms with spermicide throughout study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment emergent adverse events (TEAEs). | From baseline until the end of study (9 months)
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with adverse events of special interest (AESI). | From baseline until the end of study (9 months)
Change from baseline in vital sign parameter (blood pressure) | 9 months
Change from baseline in vital sign parameter (Heart rate) | 9 months
Change from baseline in clinical laboratory test results. | 9 months
  Number and percentage of participants with low, normal or high values and normal or abnormal examinations will be presented.
Presence of IPN10200 and BoNT-A antibodies (binding and neutralising) | From baseline until the end of study (9 months)
Change from baseline in physical examination findings. | 9 months
  Number of Participants with change in physical examination findings

SECONDARY OUTCOMES:
Change from Baseline to all post-treatment visits in Modified Ashworth scale (MAS) score in the Primary target muscle group (PTMG) | from baseline until the end of study (9 months)
  MAS is a scale to assess muscle tone in the injected muscles. The muscle tone will be rated as per grading from 0 to 4, there 0 =No increase in muscle tone and 4 =Affected part(s) rigid in flexion or extension.
Change from Baseline to post-treatment Day 29 in MAS score in the PTMG. | From baseline until post-treatment Day 29
  If PD profile of IPN10200 in dose escalation indicates a peak of effect different than Day 29, the endpoint will be modified accordingly)
Change from Baseline in MAS score in all injected muscle Groups | From baseline until the end of study (9 months)
Time to onset - time to the response to treatment (a reduction of at least one grade in the MAS score). | From baseline until the end of study (9 months)
Peak of effect - maximal decrease in the MAS score from Baseline. | From baseline until the end of study (9 months)
Time to peak - time to reach the peak of effect (maximal decrease in the MAS score from Baseline). | From baseline until the end of study (9 months)
Duration of effect - duration between time to onset and last timepoint with a response to Treatment. | From baseline until the end of study (9 months)
Response to treatment as measured by at least one grade reduction in MAS score in the PTMG from Baseline | From baseline until the end of study (9 months)
Response to treatment as measured by at least one grade reduction in MAS score in all injected muscles from Baseline | From baseline until the end of study (9 months)
Physician's Global Assessment (PGA) score of overall treatment response | From baseline until the end of study (9 months)
  The PGA is a 9-point scale (from -4= markedly worse to +4=markedly improved) used to assess global overall treatment response by the investigator.
Patient Global Impression of Change in the Spastic Clinical Pattern using specific scale (PGI-c) | from baseline until the end of study (9 months)
  PGI-C is a scale to assess global impression of change in the spastic clinical pattern using a 7-point Likert scale (from -3: very much worse to +3: very much improved) by answering a specific question
Change from Baseline in the Disability Assessment Scale (DAS) | From baseline until the end of study (9 months)
  The DAS will be used to assess the effect of upper limb spasticity on hygiene, dressing, limb position and pain. Participants will be assessed in an interview format.
Reduction of pain in the shoulder (adducted/rotated pattern) using the Numeric Rating Scale | From baseline until the end of study (9 months)
The number and percentage of participants with presence of IPN10200 and BoNT-A antibodies and titres (binding and neutralising) | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (61):
- United States (5):
  - Rancho Los Amigos National Rehab, Downey, California
  - Kansas Institute of Research, Overland Park, Kansas
  - Quest Research Institute, Farmington Hills, Michigan
  - Einstein Physical Medicine and Rehabilitation at Elkins Park, Elkins Park, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
- Austria (3):
  - Kepler University Hospital GmbH, Department of Neurology and Psychiatry, Linz
  - Brothers of Charity Hospital Linz, Department of Neurology I, Linz
  - Medical University Vienna, Department of Neurology, Vienna
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment "Heart and Brain", Pleven
  - Medical Center "Rusemed" EOOD, Rousse
  - Multiprofile Hospital for Active Treatment of Neurology and Psychiatry "Sveti Naum", Sofia, Neurological Diseases Clinic for Neurodegenerative and Peripheral Neurological Diseases, Sofia
  - Diagnostic Consulting Center - Convex EOOD, Sofia
  - Medical Center Medica Plus Ltd, Veliko Tarnovo
- Czechia (6):
  - University Hospital Hradec Kralove, Clinic of Neurology, Hradec Králové
  - Hospital Jihlava, Department of Neurology, Jihlava
  - University Hospital Ostrava, Clinic of Neurology, Center for Demyelinating diseases, Ostrava
  - Regional Hospital Pardubice, Clinic of Neurology, Pardubice
  - University Hospital Kralovske Vinohrady, Clinic of Neurology, Prague
  - General University Hospital in Prague, Clinic of Neurology, Prague
- Germany (8):
  - University Hospital Bonn, Clinic and Policlinic for Neurology, Bonn
  - Heinrich Heine University Medical Center, Department of Neurology, Düsseldorf
  - University Medicine Goettingen, Department of Neurology, Goettigen
  - University Hospital Hamburg-Eppendorf, Clinic and Polyclinic of Neurology, Hamburg
  - University Hospital Johannes Gutenberg - University of Mainz, Clinic and Polyclinic of Neurology, Mainz
  - Ludwig Maximilians University Hospital, Campus Grosshadern, Department of Neurology, Munich
  - GFO Clinics Troisdorf, St. Johannes Sieglar, Troisdorf
  - University Hospital Tuebingen, Department of Neurology, Tübingen
- Hungary (5):
  - Semmelweis University, Rehabilitation Clinic, Rehabilitation Department of Brain Injuries, Budapest
  - University of Debrecen Clinical Center, Department of Medical Rehabilitation and Physical Medicine, Debrecen
  - Petz Aladar University Teaching Hospital, Department of Neurology, Győr
  - Szent Damjan Greek Catholic Hospital, Department of Neurology and Stroke, Kisvárda
  - Borsod-Abauj-Zemplen County Central Hospital and University Educational Hospital, Department of Neurology, Miskolc
- Japan (3):
  - Fukuoka Rehabilitation Hospital, Fukuoka
  - Chutoen General Medical Center, Department of Rehabilitation, Shizuoka
  - NHO Murayama Medical Center, Department of Rehabilitation, Tokyo
- Poland (15):
  - St Wojciech - Adalbertus Hospital, Neurology Department, Gdansk
  - Specialist Doctor Practice, Katowice
  - Ma-Lek MS Therapy Centre, Katowice
  - Neuro-Medic, Katowice
  - Specialist Practises LLC, Krakow
  - Linden Medical Center, Krakow
  - Clinical Center for Neurology Sp. z o .o. (LLC), Krakow
  - NeuroKlinika - Private Practice Prof. Andrzej Bogucki, Lodz
  - Health Institute Dr n. med. Magdalena Boczarska-Jedynak, Oświęcim
  - Clinical Research Center SP. ZOO MEDIC-R, Poznan
  - Neuro-Kard Ilkowski and Partners, Poznan
  - Holy Spirit Specialist Hospital in Sandomierz - Neurology Teaching Hospital, Neurology Department, Sandomierz
  - Wolski Hospital, Neurological Department, Warsaw
  - NeuroProtect Medical Center, Warsaw
  - EuroMediCare Specialist Outpatient Clinics in Wroclaw, Wroclaw
- Russia (6):
  - Federal Siberian Research and Clinical Center, Department of Nervous Diseases, Traditional Medicine with Course in Postgraduate Education, Krasnoyarsk
  - National Medical Research Center Treatment and Rehabilitation Center, Department of Neurology, Moscow
  - "Praximed" - Diagnostic and Rehabilitation Center, Rehalibitation Department, Saint Petersburg
  - N.P. Bekhtereva Research Institute of Human Brain, Saint Petersburg
  - Astarta, LLC, Department of Neurology, Saint Petersburg
  - Medical and Sanitary Unit #70 of "Passazhiravtotrans", Saint Petersburg
- Spain (5):
  - Hospital Maritimo de Oza, A Coruña
  - University Hospital Vall d'Hebron, Barcelona
  - University Hospital de La Princesa, Physical Medicine and Rehabilitation, Madrid
  - Santiago de Compostela Clinical Hospital, Physical Medicine and Rehabilitation, Santiago de Compostela
  - Meixoeiro Hospital at Vigo University Hospital Complex, Vigo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/